CLINICAL TRIAL: NCT07293299
Title: Clinical Validation of the PneumoRator Respiratory Rate Sensor in a Perioperative Cohort
Brief Title: The PneumoRator Study
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); NIHR Southampton Respiratory Biomedical Research Centre (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0439; NIHR202107 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Respiratory; Monitored Anaesthesia Care; Perioperative
Keywords: monitoring; respiratory rate; sensor; wearable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare workers measure heart rate, blood pressure, temperature, oxygen levels and breathing rate to monitor how unwell a patient is. All these apart from breathing rate are now normally measured by machines. But there still isn't a machine that does this well enough for breathing rate to be used in most places. The machines that do exist are either uncomfortable or don't work well on patients who are moving. Instead, a healthcare worker will count the number of breaths a patient takes. This needs staff time and isn't very accurate.

It is known that changes in breathing rate can happen any time. But healthcare systems normally only measure it every few hours because it takes time. Breathing rate could be monitored all the time, we might pick up people getting sick earlier and be able to treat them more quickly, which could save lives.

A team at the University of Southampton has made a small device, called a PneumoRator, that gets stuck to onto a person's chest. Once stuck there it can measure their breathing rate and store or send that information wirelessly. The device has been tested on healthy volunteers but has never been tested on patients in hospital.

In this study the team will put the device on patients having major operations. The investigators will record information already collected about patients during normal care. This includes their breathing rate using the best measurement we have, where a patient's breathing is measured by a gas they breathe out. The gas is carbon dioxide, and the measurement is called capnography. This way of measuring is only used in operating theatres and intensive care units but is a good way to check if the PneumoRator is accurate.

The investigators want to attach the PneumoRator to patient's chests before they go to sleep for their operation and leave it there for the first few days after their operation. This will let them see how the PneumoRator compares to capnography and manual breath counting. It will also let them see how the device works at different times in the patient's journey. The investigators will look at the time when patients are asleep, when breathing is controlled by a machine. Then when patients wake up investigators can measure with both capnography and the PneumoRator. Finally, when patients go to the high dependency ward, investigators will compare it against manual counting. The study team will also ask patients how they found wearing the device and any problems they found.

With this information the investigators hope to show the PenumoRator is accurate at measuring breathing rate and comfortable for patients. This will help them get the device approved for use in hospitals and other places where breathing rate needs to be measured accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Have undergone or are referred for CPET
2. are scheduled for elective surgery and expected to have >24 hours postoperative hospital stay
3. Will be admitted to the Surgical High Dependancy Unit (SHDU) as part of their planned care
4. will receive invasive arterial pressure monitoring as part of routine care
5. are aged 18 or over
6. have the capacity to give consent to participate

Exclusion Criteria:

1. do not proceed to surgery following CPET referral
2. are aged less than 18 years
3. do not have capacity to consent
4. decline to consent
5. have sensitivity or allergy to medical adhesives
6. patients with fragile, erythematous, or broken skin at the site of PnemoRator attachment or any other condition which, in the view of the clinical research team, may mean that the use of the PnemoRator device and adhesive is likely to cause patient harm.
7. patients with implantable electronic medical devices (e.g. pacemakers, nerve stimulators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study comprises patients undergoing intermediate-high risk major surgery at University Hospital Southampton who are planned for admission to the Surgical High dependency unit (SHDU)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Agreement between respiratory rate measured by the PneumoRator device and waveform capnography | From start of anaestheisa care until departure from PACU (Recovery)

SECONDARY OUTCOMES:
Agreement between respiratory rate measured by the PneumoRator device and manual breath counting | Post-operative Day 1
Agreemement between PneumoRator and ECG based measurement of respiratory rate | Perioperatively
Patient comfort while wearing the PneumoRator | Postoperative day 1-3
  Measured using likert-scale, created specifically for this study. Higher score means more discomfort. Minimum score = 3, maximum score = 15. Questions below, (choices in brackets each rated from 1-5):
  1. How much discomfort, specifically related to the PneumoRator device, did you experience? (No discomfort, Mild discomfort, Moderate discomfort, Severe discomfort, Unbearable discomfort)
  2. How frequently did you experience discomfort, specifically related to the PneumoRator device? (Never, Rarely, Sometimes, Often, Constant)
  3. Having worn the PneumoRator device how concerned would you be about wearing the device in future? (Not concerned at all, Unconcerned, Neutral, Concerned, Very Concerned)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampon NHS Foundation Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No